CLINICAL TRIAL: NCT06143553
Title: A Randomized, Controlled Phase Ⅲ Study of Paclitaxel Polymeric Micelles for Injection Versus Physician's Choice(TPC) in Human Epidermal Growth Factor Receptor 2-negative (HER2-) Metastatic Breast Cancer (MBC) Subjects Who Have Failed at Least Two Previous Chemotherapy Regimens.
Brief Title: Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection in the Treatment of Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Yizhong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHYZ-ZSCJS-RXⅢ-01
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Breast Cancer (MBC)
Keywords: Paclitaxel Polymeric Micelles for Injection; Metastatic Breast Cancer (MBC); human epidermal growth factor receptor 2-negative (HER2-)
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; eribulin; Capecitabine; Gemcitabine; Vinorelbine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel Polymeric Micelles for Injection (Experimental): 300mg/m2 of Paclitaxel Polymeric Micelles for Injection is intravenously administrated for ≥ 3 hours without special infusion device. The frequency of administration is once every 3 weeks (Q3W), and 3 weeks constitutes a treatment cycle.
  Interventions: Drug: Paclitaxel Polymeric Micelles for Injection
- The Doctor chooses the treatment（TPC） (Active Comparator): Control Group：The Doctor chooses the treatment（TPC）：Eribulin Mesilate injection；Capecitabine Tablets；Gemcitabine Hydrochloride for Injection；Vinorelbine Tartrate Injection；Paclitaxel (albumin-bound).
  Eribulin Mesilate injection：on days 1 and 8 of the 21-day cycle, 1.4 mg/m2 , intravenous administration; Capecitabine Tablets: On days 1 to 14 of the 21-day cycle, 1000-1250mg/m2，oral administration, twice a day (once in the morning and once in the evening; Total daily dose 2000-2500mg/m2); Gemcitabine Hydrochloride for Injection: On days 1, 8 and 15 of the 28-day cycle, 800-1200mg/m2, intravenous administration; Vinorelbine Tartrate Injection: Every first day of the week, 25mg/m2，intravenous administration; Paclitaxel (albumin-bound): On day 1 of the 21-day cycle, 260mg/m2，intravenous administration for more than 30 minutes. Three weeks constituted one course of treatment.
  Interventions: Drug: Eribulin Mesilate injection; Drug: Capecitabine Tablets; Drug: Gemcitabine Hydrochloride for Injection; Drug: Vinorelbine Tartrate Injection; Drug: Paclitaxel (albumin-bound)

INTERVENTIONS:
Drug: Paclitaxel Polymeric Micelles for Injection — Subjects are given 300 mg/m2 of Paclitaxel Polymeric Micelles for Injection without special infusion device,intravenously administrated for ≥ 3 hours.Three weeks constituted one course of treatment.
  Arms: Paclitaxel Polymeric Micelles for Injection
Drug: Eribulin Mesilate injection — Subjects are given 1.4 mg/m2 of Eribulin Mesilate injection on days 1 and 8 of the 21-day cycle.
  Arms: The Doctor chooses the treatment（TPC）
Drug: Capecitabine Tablets — Subjects are given 1000-1250mg/m2 of Capecitabine Tablets on days 1 to 14 of the 21-day cycle ,and twice a day (once in the morning and once in the evening; Total daily dose 2000-2500mg/m2).
  Arms: The Doctor chooses the treatment（TPC）
Drug: Gemcitabine Hydrochloride for Injection — Subjects are given 800-1200mg/m2 of Gemcitabine Hydrochloride for Injection on days 1, 8 and 15 of the 28-day cycle.
  Arms: The Doctor chooses the treatment（TPC）
Drug: Vinorelbine Tartrate Injection — Subjects are given 25mg/m2 of Vinorelbine Tartrate Injection every first day of the week.
  Arms: The Doctor chooses the treatment（TPC）
Drug: Paclitaxel (albumin-bound) — Subjects are given 260mg/m2 of Paclitaxel (albumin-bound) on day 1 of the 21-day cycle,intravenous administration for more than 30 minutes.
  Arms: The Doctor chooses the treatment（TPC）

SUMMARY:
This multicenter, randomized, open, parallel positive control study compares the clinical efficacy and safety of paclitaxel polymeric micelles for injection with TPC in HER2- MBC subjects who have failed ≥2 to≤4 previous chemotherapy regimens.

Treatment Protocol: Subjects are randomized into paclitaxel polymeric micelles for injection group and the Physician's Choice (TPC) group by the proportion of 1:1. Randomization is stratified according to three factors: number of lines of previous treatment for metastatic disease (2 or 3/4 lines), receptor status (triple-negative, non-triple-negative), and visceral metastasis (yes/no).

Progression-free survival (PFS) is the main efficacy indicator in this study. Treatment Group: Subjects are given paclitaxel polymeric micelles for injection, three weeks constitutes one cycle of treatment.

Control Group: Physician's Choice Group, subjects are given Eribulin Mesilate injection; or capecitabine tablets; or gemcitabine hydrochloride for injection; or vinorelbine tartrate injection; or paclitaxel (albumin-bound). Three or four weeks constitutes one cycle of treatment.

If subject does not develop disease progression after 6 cycles of dosing, the subject continues treatment until disease progression (RECIST 1.1) or develops an intolerable toxicity, initiation of a new anti-cancer drug, withdrawal from the study, death, or loss of follow-up.

Superiority design is used in this study, progression-free survival (PFS) is the main efficacy indicator. Assuming α = 0.0249(unilateral, adjusted test level), power=80%, the median PFS of the treatment group is 6.0 months, the median PFS of the control group is 3.7 months, the enrollment period is 12 months, and the study period is 24 months. Using PASS (version 11.0) for calculation, a total of 152 subjects (76 in each group) are required to meet the statistical significance between the treatment group and the control group. In consideration of case expulsion, enlarged by 10%, a total of 168 subjects (84 in each group) are required.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must meet all the following criteria:

  1. Male or female 18 years and older;
  2. Understand the purpose, benefits and risks of this clinical trial, voluntarily participate in and sign the written informed consent;
  3. The Eastern Cooperative Oncology Group (ECOG)performance status is 0 or 1;
  4. Histologically or cytologically confirmed (local laboratory) HER2-metastatic breast cancer from recently acquired or newly acquired tumor biopsies from locally-relapsed or metastatic sites (HER2- is defined as a standard immunohistochemical (IHC) test result of 0 or 1+; Or the IHC test result is 2+ and the ISH test result is negative including FISH/CISH/SISH)；
  5. Archival slides or newly obtained biopsy slides from metastatic or recurrent sites are available (Note: Bone lesion biopsy is not accepted);
  6. Subjects who are refractory or relapsed after ≥2 and ≤4 prior systemic chemotherapy regimens or antibody-drug conjugates (ADC) for MBC are eligible(Subjects were eligible for inclusion if their previous chemotherapy regimen included taxanes or not; Subjects using taxanes for adjuvant or neoadjuvant chemotherapy more than 6 months after the treatment, and Subjects using taxanes for advanced-stage treatment more than 3 months after the treatment, with recurrence or metastasis are eligible.) Adjuvant or neoadjuvant chemotherapy for early-stage disease can be considered as one of the required prior chemotherapy regimens if unresectable, locally advanced, or metastatic disease develops within 12 months after completion of the regimen.( Note: Therapies for bone metastases (e.g., bisphosphonates, denosumab, etc.) are not considered prior systemic chemotherapy for advanced disease.)；
  7. Subjects are eligible to receive one the chemotherapy regimens in the TPC group；
  8. According to RECIST 1.1, subjects with measurable lesions on contrast-enhanced CT or MRI (≥10mm in the major dimension on CT or MRI scan, and ≥15mm in the minor dimension of lymph nodes); Subjects with unmeasurable skeletal lesions only are not accepted；
  9. Functions of major organs such as heart, lung, liver and kidney are basically normal；
  10. Blood routine examination meets the following criteria (No blood transfusions, blood products, granulocyte colony-stimulating factor, or other hematopoietic growth factors were used within 7 days before the blood routine test)：

      1. : White blood cell count ≥3.0x109/L; Neutrophil count ≥1.5x109/L；
      2. : Platelet count ≥100×109/L;
      3. ：Hemoglobin≥90g/L;
      4. : If subjects receive blood component transfusion (red blood cells, platelets, etc.) during the screening period, blood routine test should be performed again at an interval of 1 week to meet the above criteria before continuing screening.
  11. Blood biochemical examination must meet the following criteria:

      1. : Total bilirubin ≤1.5 times the upper limit of normal (ULN);
      2. : Aspartate Transaminase（AST）, Alanine Aminotransferase（ALT）, or Alkaline phosphatase（ALP）≤2.5 times ULN (ALT, AST, or ALP≤ 5×ULN for subjects with liver metastases, and ALP≤10×ULN for subjects with bone metastases);
      3. : Creatinine clearance (calculated using Cockcroft-Gault formula) ≥50 ml/min.
  12. Subjects have no symptoms of cardiac dysfunction (NYHA class ≤II) at baseline and no significant or clinically insignificant ECG abnormalities;
  13. Subjects have good compliance and voluntarily comply with the clinical trial protocol during the study, followed up by the investigators;
  14. All women of childbearing age, men of childbearing potential, or their spouses who have no plans to have children or donate sperm during the entire trial period and up to 6 months after the last dose of medication, or who voluntarily used effective contraception; Women of childbearing age who have a negative blood/urine pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* Subjects meet the following criteria are not eligible for inclusion:

  1. Known allergy or intolerance to either study treatment or any excipients；
  2. Previous use of antibody-drug conjugate (ADC) with anti-microtubule inhibitor as payload drug are not eligible;
  3. Primary brain tumors or central nervous system metastases (including leptomeningeal metastases), except for single brain metastases strictly controlled asymptomatic subjects; Subjects with intracranial hypertension or neuropsychiatric symptoms after treatment of central nervous system tumors;
  4. Subjects with acute or chronic infections that have not been eliminated, or subjects with other serious diseases at the same time;
  5. Subjects have other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
  6. Subjects with a known history of clinically significant active chronic obstructive pulmonary disease or other moderate to severe chronic respiratory disease within 6 months before enrollment;
  7. Subjects with active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease), clinically significant gastrointestinal (GI) bleeding, intestinal obstruction, or GI perforation within 6 months before enrollment;
  8. Subjects with active hepatitis, or liver metastasis is more than 3/4 of the whole liver;
  9. Subjects with third-space effusions (e.g., moderate-to-massive pleural effusion, moderate-to-massive pericardial effusion, ascites) that cannot be controlled by drainage or other means; Subjects with a small amount of pleural effusion without clinical symptoms and no need for clinical intervention should be strictly controlled before enrollment;
  10. Subjects with mental illness or disorder, poor compliance, or inability to cooperate, or describe treatment responses;
  11. Subjects who cannot tolerate chemotherapy due to severe organic disease or major organ failure, such as decompensated heart and lung failure;
  12. Subjects with bleeding disorders;
  13. Subjects with organ transplant;
  14. Subjects with bad drug addicts, long-term alcoholics, infectious diseases such as AIDS;
  15. Subjects on long-term use of adrenocortical hormones or immunosuppressants;
  16. Subjects who received vaccines (including live and live attenuated vaccines) such as measles, mumps, rubella, varicella, yellow fever, rabies, Bacille Calmette-Guérin vaccine（BCG ）and typhoid (oral) vaccines within 4 weeks before enrollment, or are scheduled to receive vaccines during the study period; Subjects who received all types of COVID-19 vaccines within two weeks before enrollment;
  17. Subjects who received antineoplastic drugs (including but not limited to chemotherapy, hormonal therapy, immunotherapy, antibody therapy, radiotherapy, surgery (except diagnostic biopsy), etc.) within 2 weeks before enrollment or who still have grade ≥2 toxicity from previous antineoplastic therapy (except alopecia and grade ≤2 neurotoxicity caused by platinum) at enrollment;
  18. Subjects with active hepatitis B or C (previous history of hepatitis B infection, with or without drug control, HBV DNA≥1×104 copies or ≥2000 IU/mL; Hepatitis C infection, HCV RNA≥15IU/mL); Or HIV antibody positive (testing is not necessary if there is no clinical evidence to suggest possible HIV infection);
  19. Subjects are considered not able to complete the trial or otherwise unfit to participate in the study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | Randomization to measured PD or date of death from any cause（up to 24 months)
  PFS(Progression-Free-Survival) was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurred first

SECONDARY OUTCOMES:
Objective response rate | Baseline to measured PD（up to 24 months)
  Objective response rate is defined as the proportion of subjects with complete or partial response as determined by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Overall survival | Randomization to date of death from any cause（up to 24 months)
  Overall survival was the time from randomization until the date of death from any cause. Participants who were alive at the end of the follow-up period (or lost to follow#up) were censored on the last date the participant was known to be alive.
Disease Control Rate | Baseline to measured PD（up to 24 months)
  Proportion of subjects who have achieved complete response (CR), partial response (PR) or stable disease (SD) (RECIST 1.1)
Incidence of adverse events | up to 24 months
  Safety Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Yin, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Jiong Wu, Principal Investigator — Fudan University; Jian Zhang, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Jiangsu province Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality